CLINICAL TRIAL: NCT04406064
Title: Viral Specific T-cells (VSTs) for Treatment of SARS-CoV-2/COVID-19
Brief Title: Viral Specific T-cells for Treatment of COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The use of steroids to treat COVID prevents the use of VSTs for these patients. The Principal Investigator does not feel the study had an expectation of enrolling patients as the treatment options for COVID have evolved.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Hoxworth Blood Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0353
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Viral Infection
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Viral Specific T-cells (VSTs) (Experimental)
  Interventions: Biological: Viral Specific T-cells (VSTs)

INTERVENTIONS:
Biological: Viral Specific T-cells (VSTs) — VSTs will be infused into study participants who have evidence of SARS-CoV-2 infection.

SUMMARY:
The purpose of this research study is to learn more about the use of viral specific T-lymphocytes (VSTs) when given in the presence of COVID-19 signs and symptoms, caused by the virus SARS-CoV-2. VSTs are cells specially designed to fight viral infections. These cells are created from a blood sample collected from a donor who has recovered from COVID-19 infection. VSTs are investigational meaning that they are not approved by the Food and Drug Administration (FDA).

COVID-19 is a new virus and treatment options are evolving rapidly. VSTs have been successfully used to treat many different viral infections and may be beneficial in treating COVID-19 in the absence of other treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have evidence of infection with SARS-CoV-2
2. Patients with symptomatic COVID-19 disease, as defined by at least one of the following

   1. Imaging (CXR, CT scan, etc.) with pulmonary infiltrates consistent with COVID-19 infection
   2. Requirement for supplemental oxygenation
   3. Need for additional respiratory support, including, but not limited to High flow 02, CPAP, BiPAP, Mechanical ventilation
3. Age >1 day
4. Clinical status must allow tapering of steroids to < 0.5mg/kg prednisone or other steroid equivalent
5. Have failed at least one FDA-approved treatment for COVID-19 disease
6. Must be able to receive VST infusion in Ohio (informed consent obtained by CCHMC PI or sub-investigator either in person or by phone)

Exclusion Criteria:

1. Uncontrolled bacterial or fungal infection
2. Uncontrolled relapse of malignancy
3. Unlikely to survive within 48 hours of VST infusion

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Successful production of viral specific T-cells | Within 30 days post culture initiation
  Of the patients who had a VST culture initiated, successful production of VST cells is defined as meeting the protocol-defined release criteria.

SECONDARY OUTCOMES:
Presence of viral-specific T-cells | At 30 days after infusion
  Presence of viral-specific T-cells in the participant's blood will be assessed by Elispot assay

CONTACTS AND LOCATIONS:
Overall Officials: Adam Nelson, MBBS, FRACP, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States